CLINICAL TRIAL: NCT06780631
Title: The Effect of Web-Based and Face-to-Face Education Based on the Health Promotion Model on Foot Care Behavior in Individuals With Type 2 Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Aysun Kürkçü, PhD Candidate, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 09.2023.240
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Foot; Diabetes Mellitus Type 2
Keywords: Diabetic Foot; Self Care; Health Promotiom Model; Web Based Education; Face to Face Education
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: It is a prospective intervention type three-group randomized controlled clinical study. Distribution according to the groups and layers to be assigned for each intervention; Group-1 (Experiment) was designed as web-based diabetic foot training, Group-2 (Experiment) was designed s face-to-face diabetic foot training, and Group-3 (Control) was designed as clinical routine training.
Who Masked: Outcomes Assessor
Masking Description: Due to diabetic foot training was applied as an intervention, patients and the researcher will not be considered blind. The evaluator will be considered blind in the analysis of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group-1 (Web-based diabetic foot education applied group) (Experimental): 1. In the first interview, individuals in the web training group who met the inclusion criteria and agreed to participate in the research; Within the scope of the pre-test, the Patient Information Form, Diabetic Foot Information Scale, Foot Care Behavior Scale and Diabetic Foot Care Self-Efficacy Scale will be administered by the researcher in the diabetes education unit of the hospital.
  2. After the pre-test, a username and password will be defined for individuals in the web training group so that they can log in to the diabetic foot web training page.
  3. Patients will be trained on how to access the diabetic foot web training page, how to access information, and how to use videos.
  4. After the first application, in the first and third months, patients will be invited to the diabetes education unit and the Diabetic Foot Knowledge Scale, Foot Care Behavior Scale and Diabetic Foot Care Self-Efficacy Scale will be re-administered by the researcher through face-to-face interviews.
  Interventions: Other: Web-based diabetic foot education based on health promotion model
- Group-2 (Face to face diabetic foot education applied group) (Experimental): 1. In the first meeting for individuals in the face-to-face education group; Within the scope of the pre-test, the Patient Information Form, Diabetic Foot Information Scale, Foot Care Behavior Scale and Diabetic Foot Care Self-Efficacy Scale will be administered by the researcher in the diabetes education unit of the hospital.
  2. After the pre-test, face-to-face diabetic foot training will be given in accordance with the training booklet for approximately 45 minutes.
  3. After the first application, in the first and third months, patients will be invited to the diabetes education unit and the Diabetic Foot Knowledge Scale, Foot Care Behavior Scale and Diabetic Foot Care Self-Efficacy Scale will be re-administered by the researcher through face-to-face interviews.
  Interventions: Other: Face to face diabetic foot education based on health promotion model
- Group-3 Clinical routine education applied group (control) (No Intervention): 1. In the first interview, individuals in the control group who met the inclusion criteria and agreed to participate in the research; Within the scope of the pre-test, the Patient Information Form, Foot Care Behavior Checklist, Diabetic Foot Knowledge Scale, Foot Care Behavior Scale and Diabetic Foot Care Self-Efficacy Scale will be administered by the researcher in the diabetes education unit of the hospital. 2. After the pre-test, individuals in the control group will receive routine training given by the training nurse on duty in the diabetes education unit. Education based on the health promotion model will not be implemented. 3. After the first application, in the first and third months, patients will be invited to the diabetes education unit and the Diabetic Foot Knowledge Scale, Foot Care Behavior Scale and Diabetic Foot Care Self-Efficacy Scale will be re-administered by the researcher through face-to-face interviews.

INTERVENTIONS:
Other: Web-based diabetic foot education based on health promotion model — The first group can access the training at any time and repeat the training thanks to web-based training.
  Arms: Group-1 (Web-based diabetic foot education applied group)
Other: Face to face diabetic foot education based on health promotion model — Individuals with Type 2 diabetes in the face-to-face training group will receive face-to-face diabetic foot training in line with the training booklet for approximately 45 minutes, one by one.
  Arms: Group-2 (Face to face diabetic foot education applied group)

SUMMARY:
Diabetic foot is a complication that develops difficult-to-heal foot wounds, reduces the quality of life of individuals with diabetes, causes loss of productivity, and causes economic burden due to the repetition of the problem and the expenditures made for treatment. Diabetic foot is the most common complication requiring hospitalization and is the most common cause of non-traumatic amputations. However, this complication can be prevented with regular foot examinations, patient education and daily foot care. For this reason, diabetic foot education should be given to all diabetic patients and they should be encouraged to participate in their self-care. However, educating patients once does not provide enough knowledge to manage diabetes throughout life. As the rate of individuals using web-based information increases, it is possible to reach large masses. With web-based training, information obtained from current sources is presented to patients on a single web page, patients can access training regardless of place or time, and continuity in training is ensured. The aim of this randomized controlled experimental study is to determine the effect of web-based and face-to-face education based on the health promotion model on diabetic foot knowledge and foot care behavior in individuals with diabetes.

DETAILED DESCRIPTION:
The research will be conducted with individuals with type 2 diabetes who volunteered to participate in the study. As data collection tools, Patient Descriptive Information Form, Diabetic Foot Information Scale, Foot Care Behavior Scale and Diabetic Foot Care Self-Efficacy Scale will be used. As a pre-test, data will be collected from all patients at the first interview. Then, web-based training based on the health promotion model will be applied to the individuals in the experimental group 1 and face-to-face training will be applied to the individuals in the experimental group 2. The individuals in the control group will be given routine training applied in the hospital. Reminder messages about foot care will be sent to the patients once a week. After the first application, data from all individuals in experiment group 1, experiment group 2 and control group will be collected again and analyzed in the 1st and 3rd months, and the research will be completed. Power analysis was performed using the G*Power (v3.1.9.2) program to determine the number of samples. The power of the study is expressed as 1-β (β = probability of type II error), and in general, studies must have 80% power. The number of samples was determined as 135 in total, 45 people in each group.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with type 2 diabetes at least 6 months ago according to ADA criteria
* Being between the ages of 18 and 80
* Ability to read and write
* Not having received diabetic foot training before
* No existing foot ulcers
* Using the Internet (from sources such as smartphone, tablet, computer)
* Being open to communication and collaboration
* No mental problems
* Volunteering to participate in the study

Exclusion Criteria:

* Wants to leave the study
* Foot ulcer development in a diabetic individual during work

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2024-05-17 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Diabetes Foot Knowledge Level | The knowledge level of the patients is measured with the 5-item "Diabetes Foot Knowledge Qustionnare" ; It will be evaluated before the training, in the first month and in the third month after the training.
  The scale consists of 5 items and has no subdimensions. In the evaluation of the scale, the total score of the correct questions from the answers given as 'yes' or 'no' to the knowledge question constitutes the scale score. The scoring changez as 1 or 0. An increase in the scale score indicates an increase in the level of knowledge of diabetic feet.
Foot Care Behavior | Patients' foot care behaviors will be questioned with the "Foot Self Care Observation Guide" consisting of 15 items; It will be evaluated before the training, in the first month and in the third month after the training.
  The scale consists of 15 items and has no sub-dimensions. These items are evaluated as '1=Never', '2=Occasionally', '3=Sometimes', '4=Often', '5=Always'. The lowest score on the scale is 15 and the highest score is 75. An increase in the scale score indicates that the individual's self-care behaviors are better.
Foot Care Self-Efficacy | Patients' foot care self-efficacy is evaluated with the "Diabetic Foot Care Self Efficacy" consisting of 9 items; It will be evaluated before the training, in the first month and in the third month after the training.
  The scale consists of nine items. These nine statements are evaluated on an 11-number visual scale such as 'I don't see it at all adequate = 0' and 'I consider it very adequate = 10'. The lowest score from the scale is 0 and the highest score is 90. An increase in the scale score indicates that the individual's self-efficacy is high.

CONTACTS AND LOCATIONS:
Overall Officials: Aysun Kürkçü, Principal Investigator — Kartal Dr.Lütfi Kırdar City Hospital İstanbul, Turkey
Locations (1):
- Kartal Dr.Lütfi Kırdar City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sahin S, Cingil D. Evaluation of the relationship among foot wound risk, foot self-care behaviors, and illness acceptance in patients with type 2 diabetes mellitus. Prim Care Diabetes. 2020 Oct;14(5):469-475. doi: 10.1016/j.pcd.2020.02.005. Epub 2020 Feb 27. PMID 32115378
- [Result] Pourkazemi A, Ghanbari A, Khojamli M, Balo H, Hemmati H, Jafaryparvar Z, Motamed B. Diabetic foot care: knowledge and practice. BMC Endocr Disord. 2020 Mar 20;20(1):40. doi: 10.1186/s12902-020-0512-y. PMID 32192488
- [Result] Kilic M, Karadag A. Developing and Evaluating a Mobile Foot Care Application for Persons With Diabetes Mellitus: A Randomized Pilot Study. Wound Manag Prev. 2020 Oct;66(10):29-40. PMID 33048829
- [Result] Chau JP, Chung LC, Wong RY, Loo KM, Lo SH, So TT, Lau MS, Yeung TH, Leung BS, Tong ML, Li CY, Kwok WW, Thompson DR, Lee DT. An evaluation of a web-based diabetes education program designed to enhance self-management among patients living with diabetes. Comput Inform Nurs. 2012 Dec;30(12):672-9. doi: 10.1097/NXN.0b013e318261f1d2. PMID 22872044
- [Result] Abrar EA, Yusuf S, Sjattar EL, Rachmawaty R. Development and evaluation educational videos of diabetic foot care in traditional languages to enhance knowledge of patients diagnosed with diabetes and risk for diabetic foot ulcers. Prim Care Diabetes. 2020 Apr;14(2):104-110. doi: 10.1016/j.pcd.2019.06.005. Epub 2019 Jul 13. PMID 31311727
- See also: Diabetes Foot Knowledge Qustionnare — https://tez.yok.gov.tr/UlusalTezMerkezi/TezGoster?key=EEdeQgIdFRxX5NbvVau-Agx-1m7dkjzIPn8VvT6DbLpWfi2FpSk17kl01m8WKqMg
- See also: Foot Self Care Observation Guide — https://tez.yok.gov.tr/UlusalTezMerkezi/TezGoster?key=EEdeQgIdFRxX5NbvVau-Agx-1m7dkjzIPn8VvT6DbLpWfi2FpSk17kl01m8WKqMg
- See also: Diabetic Foot Care Self Efficacy Scale — https://tez.yok.gov.tr/UlusalTezMerkezi/TezGoster?key=EEdeQgIdFRxX5NbvVau-Agx-1m7dkjzIPn8VvT6DbLpWfi2FpSk17kl01m8WKqMg